CLINICAL TRIAL: NCT06807073
Title: Complete Closure After Endoscopic Mucosal Resection of Large Non-Pedunculated Colorectal Polyps: a Randomized Controlled Trial
Brief Title: Complete Closure After Endoscopic Mucosal Resection of Large Non-Pedunculated Colorectal Polyps
Acronym: Closure-RCT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Principal Investigator, Daniel Von Renteln, Gastroenterologist, MD, Centre hospitalier de l'Université de Montréal (CHUM)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-12350
Record Dates: First submitted 2025-01-29; First posted 2025-02-04 (Actual); Last update posted 2025-02-11 (Actual); Status verified 2025-02

CONDITIONS: Colorectal Cancer; Polyp of Colon
MeSH Terms: conditions — Colorectal Neoplasms; Colonic Polyps

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endoscopic Mucosal Resection (EMR) + prophylactic defect closure (defect closure) (Experimental): Prophylactic defect closure will be performed using at least one new generation closure device.
  Interventions: Procedure: Prophylactic defect closure
- Endoscopic Mucosal Resection (EMR) (Active Comparator): After performing EMR with thermal ablation, prophylactic defect closure will not be performed.
  Interventions: Procedure: No prophylactic defect closure

INTERVENTIONS:
Procedure: Prophylactic defect closure — Endoscopists will use at least one new generation closure device to approximate the healthy mucosal surrounding the submucosal defect to ensure complete defect closure. Adequate apposition of the mucosal defect margins will be achieved when no visible submucosal areas >3 mm along the closure line are present.
  Arms: Endoscopic Mucosal Resection (EMR) + prophylactic defect closure (defect closure)
Procedure: No prophylactic defect closure — After performing EMR with thermal ablation, prophylactic defect closure will not be performed.
  Arms: Endoscopic Mucosal Resection (EMR)

SUMMARY:
The goal of this clinical trial is to compare adverse even rates after EMR for large (≥20mm) flat colorectal polyps (so-called laterally spreading lesions, LSLs) when performing complete or no defect closure. It will also evaluate lesion recurrence after EMR for large colorectal LSLs.

The hypothesis is that performing complete defect closure following EMR of large colorectal LSLs will result in lower rates of adverse events compared to cases where no defect closure is performed.

For participants with planned EMR, endoscopists will perform EMRs as per standard of care and:

* prophylactic defect closure will either not be performed (control group), or will be performed (experimental group);
* then, patients will be called between 14 and 44 days after EMR to assess for possible adverse events, and electronic medical files will be verified for emergency room visits and healthcare received for an adverse event;
* finally, patients will undergo follow-up colonoscopy 6 months and 18 months after randomization.

DETAILED DESCRIPTION:
This trial is an open-label, two-arm, parallel-group, multicenter, randomized controlled superiority trial. Patients undergoing EMR will be randomized in a 1:1 ratio and assigned to undergo no closure (control group) vs complete defect closure (experimental group).

Participants with planned EMR procedures will be approached by a research assistant before the EMR to request study participation. To mitigate loss to follow-up, patients will be questioned on their preferred contact method with multiple contact methods obtained to adequately reach patients. The importance of follow-up after EMR to detect and treat recurrence will also be highlighted both verbally and in the consent forms during initial patient contact.

Despite being experienced, all endoscopist participants will review dedicated teaching videos showing the standardized EMR approach. Videos demonstrating key technical details defect closure will also be circulated across sites to ensure a standardized approach for both procedures as described in the literature.

- Control group: EMR will be performed as per standard of care with submucosal injection and electrocautery resection of all visually visible polyp tissue using a snare. After performing EMR with thermal ablation, prophylactic defect closure will not be performed. Endoscopists can chose to close defects if there are significant concerns for risk of perforation or active perforation after EMR. When the endoscopist determines that the resection is complete, a tattoo will be placed 3 cm distal to the resected lesion to allow for better identification of the resection site in case of follow-up colonoscopy for delayed bleeding. If multiple large polyps are found and removed, the largest lesion (study polyp) will be marked with two tattoos 3 cm distal and 3 cm proximal to the lesion, to clearly identify the study polyp resection site.

- Experimental group: EMR will be performed as per standard of care with submucosal injection and electrocautery resection of all visually visible polyp tissue using a snare.

After performing EMR with thermal ablation, prophylactic defect closure will be performed. The choice of the number and types of closure devices used to achieve defect closure will be left to endoscopist discretion. If multiple large polyps are found and removed, the largest lesion (study polyp) will be marked with two tattoos 3 cm distal and 3 cm proximal to the lesion, to clearly identify the study polyp resection site. As per standard of care, endoscopists will take a photograph of the lesion before resection for documentation; a photograph of the EMR resection site will be taken before and after defect closure; a photograph of the defect will be taken if emergency colonoscopy is performed to treat delayed bleeding. When more than one lesion meeting inclusion criteria is present in a patient, all lesions 20mm or larger will be photographed next to an open snare to aid in size measurement.

- 6-month & 18-month follow-up colonoscopies: To mitigate loss to follow-up, patients will be questioned on their preferred contact method with multiple contact methods obtained to adequately reach patients. The importance of follow-up after EMR to detect and treat recurrence will also be highlighted both verbally and in the consent forms during initial patient contact. Patients will be sent a reminder that they will soon receive an invitation to undergo follow-up through their preferred contact method. If patients do not undergo follow-up after invitation, a research assistant will contact patients by phone to answer any concerns they might have at that time.

At follow-up colonoscopies, endoscopists will identify the resection scar tangential to the tattoo placed at the initial EMR. The resection scars will be observed under white light and digital chromoendoscopy to assess for visual recurrence. For all patients, four random biopsies will be taken at the resection scar. If visual recurrence is present, the lesions will be resected using the method deemed most appropriate by the endoscopist at the time and pathologically evaluated for histologic recurrence.

ELIGIBILITY:
Inclusion Criteria:

* adult ≥18 years old
* patients undergoing EMR for a large (≥20mm) colorectal LSL
* patients providing written and informed consent for study participation.

Exclusion Criteria:

* inflammatory bowel disease;
* non-elective colonoscopy;
* poor general health (American Society of Anesthesiologists classification >III);
* coagulopathy or thrombocytopenia (international normalized ratio ≥1.5 or platelets <50 x 109/L);
* pedunculated polyps (Paris class Ip, Isp);
* overt signs of deep submucosal invasive cancer (JNET 3);
* appendiceal orifice or terminal ileum invasion;
* pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 686 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Delayed bleeding | 14 days
  Defined as blood per rectum resulting in emergency room visit, unplanned hospitalization; endoscopic, radiologic, or surgical intervention.
Delayed perforation | 14 days
  Defined as endoscopic or radiologic evidence of air or luminal contents outside the gastrointestinal tract

SECONDARY OUTCOMES:
Any delayed bleeding | 14 days
  Defined as blood per rectum after the procedure
Clinically significant delayed bleeding in the proximal colon | 14 days
  Defined as proximal to the splenic flexure
Clinically significant delayed bleeding in the distal colon | 14 days
  The distal colon is defined as splenic flexure and distal
Lesion recurrence | 6 months
  Lesion recurrence at 6 months' follow-up defined by pathology-confirmed hyperplastic, serrated or adenomatous histology at the tattooed resection site

OTHER OUTCOMES:
Defect closure time | 14 days
  Time for defect closure
Technical success for complete defect closure | 6 months
  Defined as adequate apposition of the mucosal defect margins without visible submucosal areas >3 mm along the closure line
Procedure costs | 18 months
  Costs associated with procedures
Technical success of margin and/or base ablation | 18 months
  Defined as achieving a complete uninterrupted ring of circumferential margin ablation for margin ablation, and achieving 100% surface ablation of the resection base for base ablation
Colonoscopies required to achieve lesion clearance | 18 months
  Defined as no histologic recurrence at the resection scar on follow-up
EMR procedure time | During procedure
  Duration of the EMR procedure
Margin and/or base ablation time | During procedure
  Duration of the margin and/or base ablation
Loss to follow-up | 18 months
  Number of patients lost to follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier de l'Université de Montréal, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures and appendices).
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 12 months and ending 36 months following article publication.
Access Criteria: Proposals should be directed to daniel.von.renteln.med@ssss.gouv.qc.ca . To gain access, data requestors will need to sign a data access agreement